CLINICAL TRIAL: NCT01422538
Title: Evaluation of the Ulthera® System for Lifting and Tightening the Face and Neck Following Sculptra® Treatment
Brief Title: Ultherapy™ Treatment Following Sculptra® Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULT-113
Record Dates: First submitted 2011-08-22; First posted 2011-08-24 (Estimated); Results first posted 2013-08-27 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy™ treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening; Skin laxity on the face and neck.
MeSH Terms: conditions — Cutis Laxa | interventions — New-Fill

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): Subjects will receive Ulthera® System alone.
  Interventions: Device: Ulthera® System
- Group B (Active Comparator): Sculptra® only
  Interventions: Drug: Sculptra®
- Group C (Active Comparator): Sculptra® treatment followed by Ultherapy™ treatment
  Interventions: Other: Sculptra® treatment followed by Ultherapy™ treatment

INTERVENTIONS:
Device: Ulthera® System — Focused ultrasound energy delivered below the surface of the skin on the lower face.
  Other Names: Ultherapy™
  Arms: Group A
Drug: Sculptra® — Injectable filler reconstituted prior to use. Injections are administered to the lower face in a combination of cross-hatching and fanning techniques. The Sculptra is injected in two treatment sessions 6 weeks apart.
  Other Names: Poly-L-Lactic acid fillers
  Arms: Group B
Other: Sculptra® treatment followed by Ultherapy™ treatment — Sculptra® administered in 2 injection sessions 6 weeks apart, then Ultherapy™ treatment 4 months following Sculptra.
  Arms: Group C

SUMMARY:
This clinical trial will evaluate clinical outcomes associated with the non-invasive Ultherapy™ treatment to improve skin laxity and tightening following a Sculptra® treatment.

DETAILED DESCRIPTION:
This study is a prospective,single-center, randomized clinical trial. Up to thirty (30) subjects will be treated. Enrolled subjects will be assigned to one of three (3) groups. Up to 10 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 35 to 60 years.
* Subject in good health.
* Skin laxity in the lower face and neck.
* Grade 1 and 2 on the Knize Scale

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat in the face and neck.
* Excessive skin laxity on the face and neck.
* No scarring in areas to be treated.
* Any open facial wounds or lesions.
* Acne on the face.
* Patients who have a history with keloid formation or hypertropic scarring
* Patients who have a hypersensitivity to injectable poly-L-lactic acid
* Presence of a metal stent or implant in the facial area to be treated.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Burns, MD, Principal Investigator — EpiCentre Park Lane
Locations (1):
- EpiCentre Park Lane, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty subjects were assigned to three treatment groups. Subjects NOT willing to pay for Sculptra were assigned to Treatment Group A. Subjects willing to pay for Sculptra were randomly assigned to either Treatment Group B or Treatment Group C.
Pre-assignment Details: Thirty subjects were enrolled and thirty subjects were treated in the study. The first subject was treated on June 28, 2011; the last subject was treated on March 28, 2012. The last patient follow-up for the trial was September 24, 2012.
Groups:
- Group A: Subjects received Ultherapy® Treatment only.
- Group B: Subjects received Sculptra® treatment only
- Group C: Subjects received Sculptra® treatment and Ultherapy® treatment
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 10 | 10 | 10
Completed | 10 | 8 | 8
Not Completed | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Missed visit | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group A: Subjects received Ultherapy® Treatment only. Study subjects in Group A received approximately 400 lines of Ultherapy treatment (5.0PLUS Guideline followed).
- Group C: Subjects received Sculptra® treatment and Ultherapy® treatment. Study subjects in Group C received approximately 400 lines of Ultherapy treatment (5.0PLUS Guideline followed).
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Full Range); unit: years] | 47 [37 to 56] | 47 [38 to 56] | 50 [43 to 58] | 48 [37 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 8 | 25
  Male | 3 | 0 | 2 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 9 | 10 | 9 | 28
  African American/Black | 1 | 0 | 0 | 1
  Native Amer. Indian/ Alaskan Native | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
Fitzpatrick Skin Type [Number; unit: participants] — Skin Type I = White;very fair,red or blonde hair blue eyes;freckles;Always burns, never tans
  Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes;Usually burns, tans with difficulty
  Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans
  Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease
  Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily
  Skin Type VI = Black; Never burns, tans very easily
  participants
    Type 1 | 0 | 0 | 1 | 1
    Type II | 4 | 6 | 6 | 16
    Type III | 5 | 4 | 3 | 12
    Type IV | 0 | 0 | 0 | 0
    Type V | 0 | 0 | 0 | 0
    Type VI | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Lifting and Tightening of Skin as Determined by Masked Assessment of Pre- and Post-treatment Photographs.
Description: Three masked assessors reviewed pre- and 90 days post-treatment photos from 29 subjects who returned for their 90-day follow-up visit, assessing for improvement in skin laxity at 90 days post-treatment compared to baseline, i.e., lifted and tightened skin in the areas treated with the assigned study treatment based on the assigned study arm.
Time Frame: 90 days post-treatment
Measure: Number; unit: percentage of participants improved
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 10 | 10 | 9
percentage of participants improved | 40 | 30 | 33

2. Secondary Outcome: Overall Aesthetic Improvement at 90 Days Post-treatment
Description: At 90 days post-treatment, each site investigator and each subject completed a Global Aesthetic Improvement Scale (GAIS) (Physician GAIS - PGAIS; Subject GAIS - SGAIS), comparing to pre-treatment photos. The GAIS is 5-point scale (1-5) describing an overall assessment as follows:
  1. = Very Much Improved
  2. = Much Improved
  3. = Improved
  4. = No Change
  5. = Worse "Any Improvement" includes subjects assessed in categories 1-3.
Time Frame: 90 days post-treatment.
Measure: Number; unit: percentage of participants improved
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 10 | 10 | 9
percentage of participants improved
  PGAIS - Improved to Very Much Improved | 50 | 60 | 67
  SGAIS - Improved to Very Much Improved | 70 | 60 | 56

3. Secondary Outcome: Overall Aesthetic Improvement at 180 Days Post-treatment
Description: At 180 days post-treatment, each site investigator and each subject completed a Global Aesthetic Improvement Scale (GAIS) (Physician GAIS - PGAIS; Subject GAIS - SGAIS), comparing to pre-treatment photos. The GAIS is 5-point scale (1-5) describing an overall assessment as follows:
  1. = Very Much Improved
  2. = Much Improved
  3. = Improved
  4. = No Change
  5. = Worse "Any Improvement" includes subjects assessed in categories 1-3.
Time Frame: 180 days post-treatment
Measure: Number; unit: percentage of participants improved
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 10 | 9 | 7
percentage of participants improved
  PGAIS - Improved to Very Much Improved | 30 | 33 | 43
  SGAIS - Improved to Very Much Improved | 70 | 44 | 43

4. Other Pre Specified Outcome: Subject's Assessment of Pain
Description: Subjects' sensory response to the Ulthera treatment exposures were recorded for each anatomical region treated using a validated Numeric Rating Scale (0-10), with 1 representing no pain and 10 representing the worst pain possible. Pain assessment data were obtained from Group A and Group C subjects only.
Time Frame: During Ulthera study treatment
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Group C: Subjects received Sculptra® and Ultherapy® Treatment.
Arm/Group | Group A | Group C
Number analyzed (Participants) | 10 | 10
units on a scale
  Cheek | 4.5 [2 to 8] | 4.5 [0 to 8]
  Submental | 2.9 [1 to 5] | 2.9 [0 to 6]
  Submandibular | 3.9 [1 to 7] | 3.3 [0 to 6]

5. Secondary Outcome: Subject Satisfaction at 90 Days Post-treatment
Description: Subjects rated their satisfaction as Very Satisfied, Satisfied, Dissatisfied or Very Dissatisfied using a Patient Satisfaction Questionnaire (PSQ). Responses at 90 days post-treatment Responses were tabulated.
Time Frame: 90 days post-treatment.
Population: Data analyzed includes PSQ responses at 90 days post-treatment assessing subjects' satisfaction with study treatment. Responses were tabulated. Outcomes reported represent the percentage of subjects reporting any satisfaction, i.e., Very Satisfied or Satisfied.
Measure: Number; unit: percentage of participants Satisfied
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 10 | 10 | 9
percentage of participants Satisfied | 70 | 60 | 78

6. Secondary Outcome: Subject Satisfaction at 180 Days Post-treatment
Description: Subjects rated their satisfaction as Very Satisfied, Satisfied, Dissatisfied or Very Dissatisfied using a Patient Satisfaction Questionnaire (PSQ). Responses at 180 days post-treatment Responses were tabulated.
Time Frame: 180 days post-treatment
Population: Data analyzed includes PSQ responses at 180 days post-treatment assessing subjects' satisfaction with study treatment. Responses were tabulated. Outcomes reported represent the percentage of subjects reporting any satisfaction, i.e., Very Satisfied and Satisfied.
Measure: Number; unit: percentage of participants Satisfied
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 10 | 8 | 8
percentage of participants Satisfied | 70 | 63 | 38

ADVERSE EVENTS:
Groups:
- Group B: Subjects received Sculptra® only.
Arm/Group | Group A | Group B | Group C
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
* Entrance criteria possibly restricted to a population with too little skin laxity to assess a difference.
* Group C time from Sculptra to Ultherapy may be too long to discern any added benefit of both treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No